CLINICAL TRIAL: NCT06142994
Title: Phase 4, Efficacy and Safety of Atusin CAP in the Treatment of Subjects With Acute Bronchitis in the Primary Healthcare Setting: Prospective, Multicenter, Double-blind, Placebo-controlled, Randomized, Parallel-arm Clinical Study.
Brief Title: Treatment of Adults With Acute Bronchitis in the Primary Healthcare Setting
Acronym: AАBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neopharm Bulgaria Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AАBA 2401-001
Record Dates: First submitted 2023-11-08; First posted 2023-11-22 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2023-11

CONDITIONS: Acute Bronchitis
Keywords: Cough; Sputum; Mix of essential oils; Bromelain; Green Brazilian propolis; Acute Bronchitis; Adults
MeSH Terms: conditions — Bronchitis; Cough

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, double-blind, placebo-controlled, randomized, parallel-arm clinical study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators will be provided with coded and identical products. Each individual involved in the study will be blinded to the assignment until study completion. Considering the established safety profile, emergency unblinding of treatment assignment will not be necessary, and no copies of the treatment assignments will be stored at the enrollment sites. If needed, the Investigators may receive information about the assignment of a particular subject only after review and approval by the Medical monitor. No information about the subjects will be shared with the company conducting the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum group (Experimental): 10 days of treatment with 3 daily doses of 420 mg (available in an capsule of 210 mg), as recommended by the manufacturer.
  6 capsules daily for 10 days: 2 capsules in the morning (30 minutes before breakfast), 2 capsules at noon (30 minutes before lunch), 2 capsules in the evening (30 minutes before dinner)
  Interventions: Dietary Supplement: Atusin CAP
- Placebo (Placebo Comparator): 10 days treatment with a 3-day dose of 420 mg placebo capsules (available in an indistinguishable capsule of 210 mg).
  6 capsules daily for 10 days: 2 capsules in the morning (30 minutes before breakfast), 2 capsules at noon (30 minutes before lunch), 2 capsules in the evening (30 minutes before dinner)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Atusin CAP — This food supplement contains a distillate of 4 types of purified oils - eucalyptus, sweet orange, lemon and myrtle, rich in 1,8-cineol, limonene, alpha-pinene in the ratio: 66:32:1:1, bromelain and green Brazilian propolis in a gastro-resistant capsule. The product contains excipients: microcrystalline cellulose, silica dioxide, copovidone, magnesium stearate.
  Arms: Verum group
Dietary Supplement: Placebo — The placebo product will be identical in shape, appearance and color to the active product and will have the same composition but without the active ingredients.
  Arms: Placebo

SUMMARY:
The study aims to evaluate the effectiveness and safety of Atusin® CAP in reducing the severity of acute bronchitis.

DETAILED DESCRIPTION:
A prospective, multicenter, double-blind, placebo-controlled, randomized, parallel study will be conducted to evaluate the effect of Atusin® CAP on the rapid relief of irritating cough in adults with acute bronchitis treated in actual clinical practices in primary healthcare, where patients seek help as a result of serious complaints.

The combination of the three extracts: a mix of essential oils, bromelain and green Brazilian propolis may represent a breakthrough in symptomatic treatment by blocking the triggering mechanisms of cough due to acute bronchitis.

ELIGIBILITY:
Inclusion Criteria:

Male and female ambulatory subjects

1. Age of 18 to 60 years
2. Clinical diagnosis of "Acute bronchitis" meeting the following criteria:

   * ≥6 cough attacks in the day preceding the screening visit;
   * Bronchitis Severity Scale (BSS) ≥ 5 point at screening (out of 20 points maximum);
   * Cough severity of ≥4 on the Visual Analogue Scale (VAS) at screening
   * Body temperature < 39.0°C
3. Duration of symptoms ≤ 5 days before enrollment in the study;
4. Occurrence of initial symptoms (sputum production with impaired expectoration) within 2 days prior to initiation of study treatment;
5. Good physical and mental condition;
6. Non-smokers (Active smoking of < 5 cigarettes per day or subjects who stopped smoking at least six months before enrollment in the study).
7. BMI: 18,0 - 29,9 kg/m2
8. In the judgement of the Investigator, the subject is capable of adhere with the visit schedule, complying with study treatment regimen and completing the study.
9. The subject has a smartphone and is capable of using it.
10. The subject must sign an informed consent form approved by an Ethics Committee and must agree to carry out the necessary visits to the site.

Exclusion Criteria:

1. History of or current confounding respiratory disease (for example, COPD, allergic rhinitis, chronic sinusitis or chronic bronchitis - including acute exacerbations, emphysema, bronchiectasias, asthma, cystic fibrosis, tuberculosis, lung cancer, etc.); lung radiogram revealing pulmonary inflammatory lesions; suspected pneumonia - imaging diagnostics is used mainly to rule out pneumonia.

   ACCP 2006 Guidelines point out that an imaging assessment is not indicated in patients with symptoms of acute bronchitis, who have normal vital signs and normal pulmonary evaluation.33 Absence of the following findings reduces the likelihood of pneumonia sufficiently to eliminate the need of chest radiogram or hospital admission:
   * heart rate > 100 beats/min;
   * respiratory rate > 24 breaths/min;
   * oral body temperature > 39,0 C;
   * blood pressure: systolic < 90 mmHg, diastolic < 60 mmHg;
   * SaO2 < 92%; If Investigator suspect pneumonia, the subject will not be enrolled in the study until the diagnosis of "Pneumonia" is ruled out;
2. Concurrent bacterial infection;
3. Elevated body temperature (> 39,5°C rectal or ≥39,0°C axillary);
4. Subject administers antibiotics at the time of screening or for whom antibiotics are indicated, in the judgment of the Investigator;
5. History of cough lasting over 5 days;
6. Active smoking of ≥ 5 cigarettes per day;
7. Hypersensitivity to the study treatment;
8. Active concurrent disease which may interfere with subject's ability to participate in the study, in the judgement of Investigator:

   * Sleep apnea;
   * Elevated liver enzymes (≥ 3 times the upper limit of normal (ULN));
   * Severe kidney dysfunction (glomerular filtration rate < 30 mL/min);
   * Uncontrolled diabetes mellitus (plasma glucose ≥ 250 mg/dL);
   * Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg);
   * Active peptic ulcer and gastrointestinal bleeding; coagulopathy; cataract(s); advanced malignant disease; significant cardiac disease (for example heart failure class III/IV, pulmonary hypertension, peripheral artery disease);
9. Antibiotics, antivirals, steroids, anticoagulants; treatment with antitussives or expectorants in the 7 days prior to enrollment in the study; monoamine oxidase (MAO) inhibitors (for example, antidepressants, antipsychotics, or medications for Parkinson's disease) within 2 weeks prior to randomization;
10. Subjects in poor condition requiring urgent hospitalization, or planned hospitalization during the study;
11. Women who are pregnant or lactating;
12. Women who plan on getting pregnant during the study;
13. Participation in a clinical study within the last 8 weeks;
14. Evidence or suspicion of non-compliance;;
15. Risk of lost to follow-up;
16. Inability to give informed consent;
17. Alcohol or drug abuse in the last year;
18. Unstable medical conditions, as determined by the Investigator;
19. Inability to comply with the study protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 310 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Bronchitis severity assessment | Up to 14+2 days after starting treatment
  The bronchitis severity assessment will be performed using the Bronchitis Severity Scale by the Investigator. The intensity of symptoms - frequency of coughing attacks, sputum discharge, rales on auscultation, chest pain on coughing and dyspnea will be assessed using a 5-point Likert scale: 0=Absent (1-2 times/day), 1=mild (3-5 times/day), 2=moderate (6-10 times/day), 3=severe (11-20 times/day), 4=very severe (>20 times/day).
  Clinical cure is defined as ⩾75% reduction in baseline Bronchitis Severity Scale after 10 days.

SECONDARY OUTCOMES:
Reduction in cough severity | Up to 14+2 days after starting treatment
  The severity of the cough by Visual Analogue Scale (VAS) is a single element measure of the subject's current perception of the severity of the cough. It is rated on a scale of 10 cm (100 mm), where "0" stands for "Absent" and "10" represents "The most severe possible cough".
  The decrease in cough severity per VAS by ⩾ 20 mm is assumed to be significant in this study.
Reduction of the duration (in days) of moderate to severe cough | up to 14+2 days after start of treatment
  Number of continuous days with moderate to severe cough. The severity of cough is assessed by the subject every evening at bedtime on Day 1 through Day 10, using the Visual Analogue Scale (VAS). The duration of moderate to severe cough will be calculated taking into account the number of consecutive days (2, 3,..10) in which the subject noted severity of cough of ≥ 5.
Frequency of daytime cough attacks | Up to 14+2 days after start of treatment
  An attack is defined as a single cough of 3 or more consecutive coughs. Evaluated by:
  * Investigator at subject enrollment, during screening at Visit 1 (V1) (Day 1), and the data will serve as a baseline, and on V2, V3 and V4 using the Bronchitis Severity Scale.
  * Subject every evening at bedtime on Day 1 through Day 10, using an Acute Bronchitis Severity Score.
Reduction in the frequency of nocturnal cough | Up to 10 days after the start of treatment
  The baseline frequency of cough attacks is evaluated by the Investigator at subject enrollment during screening Visit 1 (V1; CRF record) Day 1, using the Bronchitis Severity Scale and by the subject every evening at bedtime on Day 1 through Day 10, using the Acute Bronchitis Severity Score.
  The frequency of nighttime cough will be assessed daily from Day 1 (enrollment) to Day 10 and changes in its frequency will be analyzed after 1-10 days from baseline (change in day/night cough frequency after k days of treatment = frequency of day/night cough after k days of treatment - frequency of cough at enrollment (Day 1), where k = 1, 2,…,10).
Quality of life (QoL) | Up to 10 days after start of treatment
  Limitation of daily activity is assessed by the Investigator at trial entry and by subject every evening at bedtime on Day 1 through Day 10 using the Acute Bronchitis Severity Score (ABSS).
Adverse events | Up to 14+2 days after starting treatment
  Incidence of mild (e.g. self-resolving), moderate (e.g. those requiring medical evaluation) and severe (e.g. those requiring prolonged hospitalization) serious and non-serious adverse events.. Recorded daily by the subjects in ePD and by Investigators in eCRF
Response to treatment | Up to 14+2 days after starting treatment
  At each visit during/after treatment (V2, V3 and V4), response to treatment is assessed by the Investigator using a verbal rating scale (VRS): 0 = symptoms resolved [resolved], 1 = symptoms improved compared to baseline, 2 = symptoms unchanged compared to baseline, 3 = symptoms worsened compared to baseline. Subjects with points 0 or 1 are defined as "responders"; subjects with points 2 or 3 were defined as "non-responders".

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Hodzhev, Prof, PhD, Principal Investigator — Head of Pulmonology clinic in the UMHAT "Sveti Georgi", Medical University-Plovdiv; Diana Petkova, Prof, PhD, Principal Investigator — Clnic of Pneumology at UMHAT "St. Marina", Medical University - Varna; Rossen Petkov, Prof, PhD, Principal Investigator — Head of Pulmonology clinic in the UMHAT St Ivan Rilski, Medical University of Sofia; Yavor Ivanov, Prof, PhD, Principal Investigator — Head of Pneumology and Phthisiology clinic in the UMHAT "Dr. Georgi Stranski"
Locations (1):
- University Hospital "St George", Plovdiv, Bulgaria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clark TW, Medina MJ, Batham S, Curran MD, Parmar S, Nicholson KG. Adults hospitalised with acute respiratory illness rarely have detectable bacteria in the absence of COPD or pneumonia; viral infection predominates in a large prospective UK sample. J Infect. 2014 Nov;69(5):507-15. doi: 10.1016/j.jinf.2014.07.023. Epub 2014 Aug 6. PMID 25108123
- [Background] Gonzales R, Sande MA. Uncomplicated acute bronchitis. Ann Intern Med. 2000 Dec 19;133(12):981-91. doi: 10.7326/0003-4819-133-12-200012190-00014. PMID 11119400
- [Background] Braman SS. Chronic cough due to acute bronchitis: ACCP evidence-based clinical practice guidelines. Chest. 2006 Jan;129(1 Suppl):95S-103S. doi: 10.1378/chest.129.1_suppl.95S. PMID 16428698
- [Background] Tobin EH, Thomas M, Bomar PA. Upper Respiratory Tract Infections With Focus on The Common Cold. 2025 May 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK532961/ PMID 30422556
- [Background] Tackett KL, Atkins A. Evidence-based acute bronchitis therapy. J Pharm Pract. 2012 Dec;25(6):586-90. doi: 10.1177/0897190012460826. Epub 2012 Oct 16. PMID 23076965
- [Background] Malesker MA, Callahan-Lyon P, Ireland B, Irwin RS; CHEST Expert Cough Panel. Pharmacologic and Nonpharmacologic Treatment for Acute Cough Associated With the Common Cold: CHEST Expert Panel Report. Chest. 2017 Nov;152(5):1021-1037. doi: 10.1016/j.chest.2017.08.009. Epub 2017 Aug 22. PMID 28837801
- [Background] Bagcchi S. Stigma during the COVID-19 pandemic. Lancet Infect Dis. 2020 Jul;20(7):782. doi: 10.1016/S1473-3099(20)30498-9. No abstract available. PMID 32592670
- [Derived] Petkova D, Petkov R, Hodzhev V, Ivanov Y, Hadjiev V. Efficacy and safety of Atusin(R) CAP in the treatment of acute uncomplicated bronchitis in the primary care setting: a multi-center, randomized, double-blind, placebo-controlled study (AABA). BMC Pulm Med. 2025 Oct 1;25(1):443. doi: 10.1186/s12890-025-03912-6. PMID 41034950